CLINICAL TRIAL: NCT04948190
Title: Using Medical-detection Dogs to Identify People With SARS-CoV-2. Phase 2 and 3 -Training Dogs to Detect People Infected With SARS-CoV-2.
Brief Title: Canine COVID-19 Detection Phase 2 and 3
Acronym: LSH1394
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ARCTEC (Industry)
Collaborators: Durham University (Other); Cardiff University (Other); Medical Detection Dogs (Unknown)
Responsible Party: Sponsor
Other Study IDs: LSH1394
Record Dates: First submitted 2021-06-28; First posted 2021-07-01 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Covid19; SARS-CoV2 Infection
Keywords: Medical Detection Dog; Canine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Odour swab samples may be collected and retained as part of this study. These samples will comprise human sweat, and will not be used for DNA analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SARS-CoV-2 Infected/ positive group: Has tested positive for SARS-CoV-2 within appropriate timeframe (criteria vary for different study stages). Aged 16 years or older, willing and able to provide informed consent.
  Interventions: Behavioral: Testing with medical detection dogs
- SARS-CoV-2 negative group: Has tested negative for SARS-CoV-2 within appropriate timeframe (criteria vary for different study stages, and in phase 2 part 1, 2 and 4 enrolment may be accepted using symptoms-based criteria). Aged 16 years or older, willing and able to provide informed consent.
  Interventions: Behavioral: Testing with medical detection dogs

INTERVENTIONS:
Behavioral: Testing with medical detection dogs — Participants will be screened by medical detection dogs. In phase 2, participants may be asked to wear clothing samples collected in phase 1, as part of dog training procedures. In subsequent study parts, participants will wear their own clothing.

SUMMARY:
The purpose of this study is to determine whether trained medical detection dogs can accurately detect the presence of COVID-19 in people infected with the virus, or using samples of their clothing or body odour.

The study will train dogs to identify and discriminate between individuals wearing clothing collected from people infected with SARS-CoV-2 and uninfected individuals under semi-field conditions.Following this training, field testing will be used to determine whether trained dogs can distinguish between people infected with SARS-CoV-2 and uninfected individuals, producing estimates of dogs' sensitivity and specificity.

DETAILED DESCRIPTION:
When the COVID-19 epidemic wanes it will be important to prevent outbreaks of, and the reintroduction of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) into the country, since there will be many susceptible individuals remaining in the population. In order to prevent third and further waves of COVID-19, it will be important to screen passengers arriving from high-risk countries. This task would be made simpler if a rapid non-invasive method were available for detecting infected individuals, particularly those with asymptomatic, pre-symptomatic or prodromal symptomatic infections with SARS-CoV-2 from those individuals who are not carrying the virus.

Thermal screening, practised in many airports and ports around the world, has a low sensitivity since not all patients develop fever. Consequently, it has received considerable criticism in some quarters. The use of trained dogs could provide a rapid primary screen for detecting those potentially carrying the SARS-CoV-2 virus. Travellers indicated by the dogs as likely to be carrying the virus would then be tested by nasal and throat swabs, with diagnosis confirmed/excluded using real-time RT-PCR or an accurate rapid diagnostic test according to Government Guidelines. Using trained dogs would enable extremely rapid screening, with each dog able to assess up to 250 travellers per hour, saving time and money.

There is evidence that viral and bacterial respiratory infections cause the release of specific odours from human cells. Other work with detection dogs has found dogs can detect and learn the smell of virus-associated volatiles in real time, with sensitivities of up to 96% and specificity of up to 98%. The current study will build further investigate whether trained dogs can differentiate between odours associated with viral infections.

In Phase 1 of this study (Clinical Trials ref: NCT04509713), the investigators hypothesised that dogs, with their highly advanced sense of smell could be trained to detect people infected with the SARS-CoV-2 virus. Medical Detection Dogs were trained and tested using stand trials with clothing samples worn by people who had variously tested positive or negative for SARS-CoV-2 in RT-PCR tests.

In Phase 2, the clothing collected in Phase 1 will be used to train and transition the dogs from Phase 1, where they identified samples in the laboratory environment, to semi-field settings. Phase 1 clothing samples will be worn by human volunteers in a series of 'line-up' trials, under increasingly complex settings. As part of phase 2, study staff will opportunistically conduct line-up tests with volunteers confirmed to be infected with SARS-CoV-2, to allow dogs to learn the whole-body odour of infection.

Phase 3 will take place once the investigators have demonstrated the dogs can work within a real-world environment (Phase 2 above). In this phase, trainers will deploy the dogs and evaluate performance through in use testing. This will be done at a suitable venue, most likely a COVID-19 testing centre, airport or university, to ensure a high enough rate of potential positive individuals.

ELIGIBILITY:
Inclusion Criteria:

Phase 2, training part 1 & 2

* Adult male or female, aged 16 years or over.
* Written (hard copy or electronic) or verbal informed consent provided.
* Willing and able to wear or carry clothing (e.g. t-shirt) collected as part of Phase 1 from an individual infected with SARS-CoV-2 or an individual not infected with SARS-CoV-2.
* Has declared non-symptomatic 7 days (as defined by the latest NHS guidance) prior to participation in the training exercise.
* Would be willing to have a SARS-CoV-2 test within 24 h of the training exercise if required.

Phase 2, training part 3

* Adult male or female, aged 16 years or over.
* Written (hard copy or electronic) or verbal informed consent provided.
* Has received a positive result for SARS-CoV-2 from a test conducted within the past 5 days. or is experiencing SARS-CoV-2 symptoms.
* Willing and able to share, or grant access to, their SARS-CoV-2 test result.
* Has access to private outdoor space (e.g. front garden, driveway), reachable without leaving the location where the participant is self-isolating.
* Is asymptomatic or mildly ill (i.e. not requiring hospitalisation, able to walk short distances and stand for up to 15 minutes).

Phase 2 part 4, acceptability and feasibility study

* Adult male or female, aged 16 years or over.
* Written (hard copy or electronic) or verbal informed consent provided.
* Would be willing to have a SARS-CoV-2 test within 72 hours of the training exercise if required.
* Willing and able to share, or grant access to their SARS-CoV-2 test result.

Phase 2 part 5, Criteria for all volunteers

* Adult male or female, aged 16 years or over
* Electronic informed consent provided

Additional criteria for volunteers participating in focus groups

* Adult male or female, aged 16 years or over.
* Written (hard copy or electronic) or verbal informed consent provided.
* Able to access online video-conferencing tools (such as Zoom or Teams).

Phase 3, Deployment testing

* Adult male or female, aged 16 years or over.
* Willing and able to have a SARS-CoV-2 test within 96 h of participation in the deployment exercise.
* Willing and able to share, or grant access to, their SARS-CoV-2 test result.
* Verbal or written (hard copy or electronic) informed consent provided by the participant.

Exclusion Criteria:

Phase 2, training part 1 & 2

* Younger than 16 years old
* Informed consent not provided
* Unwilling or unable to wear or carry clothing from an individual infected or uninfected with SARS-CoV-2.
* Has not declared non-symptomatic within 7 days prior to the training exercise.
* Is unwilling or unable to have a SARS-CoV-2 test within 24 hours of the training exercise if required.

Phase 2, training part 3

* Adult male or female, aged under 16 years.
* Informed consent not provided.
* Has not received a positive result for SARS-CoV-2 or experiencing SARS-CoV-2 symptoms.
* Unwilling or unable to share, or grant access to their SARS-CoV-2 test result.
* Has no access to private outdoor space.
* Participant requires hospitalisation or is unable to walk short distances and stand for up to 15 minutes.

Phase 2 part 4, acceptability and feasibility study

* Adult male or female, aged under 16 years.
* Informed consent not provided.
* Unwilling or unable to have a SARS-CoV-2 test within 72 hours of the training exercise if required.
* Unwilling or unable to share, or grant access to their SARS-CoV-2 test result. Phase 2 part 5 Criteria for all volunteers
* Adult male or female, aged under 16 years.
* Informed consent not provided Additional criteria for volunteers participating in focus groups.
* Adult male or female, aged under 16 years · Informed consent not provided.
* Unable to access online video-conferencing tools (such as Zoom or Teams)

Phase 3 Deployment testing

* Adult male or female, aged under 16 years
* Informed consent not provided.
* Unwilling or unable to have a SARS-CoV-2 test within 96 hours of participation in the deployment exercise.
* Unwilling or unable to provide a scent swab.
* Unwilling or unable to share, or grant access to, their SARS-CoV-2 test result.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Phase 2 parts 1 and 2: Study population will comprise SARS-CoV-2 negative volunteers.
  Phase 2 part 3: Study population will comprise SARS-CoV-2 positive volunteers living locally to Milton Keynes.
  Phase 2 part 4: Study population will comprise attendees or passengers at relevant field location.
  Phase 2 part 5: Study population will consist of stakeholders appropriate to the field location used in phase 2 part 4.
  Phase 3: Volunteers who are seeking testing for COVID-19, or who have been tested in the past 4 days.
Sampling Method: Non-Probability Sample
Enrollment: 11015 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-09-27 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Sensitivity of dogs detecting COVID-19 on worn clothing samples. | 6 weeks
  The phase 2 study section is designed to measure the sensitivity of the dogs to detect participants infected with SARS-CoV-2 using clothing samples.
  During testing the reaction of each dog to a positive sample will be observed (i.e. standing, sitting or lying down). The dog's diagnostic accuracy will then be determined in a double-blinded study. Here the trainer and technician using the computer to record the results of the study are blinded to the identity of each sample until the trainer calls the final decision (positive or negative) based on the response of the dog to the sample.
  This outcome will assess dogs' sensitivity in screening clothing samples collected in an earlier trial, and worn by volunteers, all of whom are expected to be SARS-CoV-2 negative.
  Sensitivity will be calculated against 'gold standard' of RT-PCR test outcomes.
Phase 2: Specificity of dogs detecting COVID-19 on worn clothing samples. | 6 weeks
  The phase 2 study section is designed to measure the specificity of the dogs to detect participants infected with SARS-CoV-2 using clothing samples.
  During testing the reaction of each dog to a positive sample will be observed (i.e. standing, sitting or lying down). The dog's diagnostic accuracy will then be determined in a double-blinded study. Here the trainer and technician using the computer to record the results of the study are blinded to the identity of each sample until the trainer calls the final decision (positive or negative) based on the response of the dog to the sample.
  This outcome will assess dogs' specificity in screening clothing samples collected in an earlier trial, and worn by volunteers, all of whom are expected to be SARS-CoV-2 negative.
  Specificity will be calculated against 'gold standard' of RT-PCR test outcomes.
Phase 3: Specificity precision of dogs to detect COVID-19 in humans in semi-field settings. | 20 weeks (overlapping with phase 2)
  The phase 3 study section will measure the sensitivity of the dogs in detection of SARS-CoV-2 on human participants in semi-field settings.
  During screening the reaction of each dog to an individual being screened will be observed (i.e. standing, sitting or lying down).
  The dog's diagnostic sensitivity will be calculated by comparing these indications against outcomes of RT-PCR tests, which must be conducted within 96 hours of test participation. Testing will be conducted under double-blinded conditions.
  This outcome will assess dogs' sensitivity on in-person volunteers, screened in semi-field settings. Volunteers will comprise both SARS-CoV-2 positive and SARS-CoV-2 negative individuals.
  Sensitivity will be calculated to +/- 5% accuracy. Sensitivity= percentage of true positives correctly identified by dogs.
Phase 3: Specificity precision of dogs to detect COVID-19 in humans in semi-field settings. | 20 weeks (overlapping with phase 2)
  The phase 3 study section will measure the specificity of the dogs in detection of SARS-CoV-2 on human participants in semi-field settings.
  During screening the reaction of each dog to an individual being screened will be observed (i.e. standing, sitting or lying down).
  The dog's diagnostic specificity will be calculated by comparing these indications against outcomes of RT-PCR tests, which must be conducted within 96 hours of test participation. Testing will be conducted under double-blinded conditions.
  This outcome will assess dogs' specificity on in-person volunteers, screened in semi-field settings. Volunteers will comprise both SARS-CoV-2 positive and SARS-CoV-2 negative individuals.
  Specificity will be calculated to +/- 5% accuracy. Specificity= percentage of true negatives correctly identified by dogs.

SECONDARY OUTCOMES:
Qualitative outcome: acceptability of dogs as a screening tool | 8 weeks
  Interviews and focus groups involving stakeholder groups will be used to assess acceptability of dogs as a disease-screening tool.
  Eligible volunteers belonging to relevant groups will be invited to a single event (either interview with researcher, or focus group with other volunteers from same group type). Concept of dogs as a screening tool will be explained, using verbal overview, and where possible photos or videos.
  Volunteers will be asked to share their views on acceptability of dogs as a screening tool. Key quotes will be noted from each session. At the conclusion of all sessions, key themes and opinions will be drawn from session notes, and reported using illustrative quotes where appropriate.

CONTACTS AND LOCATIONS:
Locations (1):
- Arctec at London School of Hygiene & Tropical Medicine, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No